CLINICAL TRIAL: NCT04022005
Title: Chidamide Combined With R-GemOx(Rituximab、Gemcitabine Plus Oxaliplatin) Regimen as Salvage Treatment for Transplant-ineligible Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma: a Multi-center, Single Arm, Phase II Study
Brief Title: Chidamide + R-GemOx Regimen as Salvage Treatment for Transplant-ineligible Patients With Relapsed/Refractory DLBCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2019-091
Record Dates: First submitted 2019-07-13; First posted 2019-07-16 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Rituximab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide combined with R-GemOx (Experimental): Chidamide, 20 mg,twice per week; Rituximab 375mg/m2, d1, intravenous drip; Gemcitabine 1000mg/m2, d2, intravenous drip; Oxaliplatin 100mg/m2, d2,intravenous drip; All patients received up to 6 treatment cycles of 21 days. Patients with CR or PR will receive chidamide maintenance therapy.
  Interventions: Drug: Chidamide, Rituximab, Gemcitabine,Oxaliplatin

INTERVENTIONS:
Drug: Chidamide, Rituximab, Gemcitabine,Oxaliplatin — All patients enrolled in the study will accept Chidamide + R-GemOx (Rituximab, Gemcitabine and Oxaliplatin) as their salvage chemotherapy.
  Patients with CR or PR will receive chidamide maintenance therapy.

SUMMARY:
The purpose of this multi-center,single arm,phase Ⅱ clinical trail is to determine the safety and efficacy of Chidamide with R-GemOx(rituximab、gemcitabine plus oxaliplatin) regimen in the treatment of transplant-ineligible patients with relapsed/refractory diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proved CD20+ DLBCL;
* relapse or refractory DLBCL#
* previously received systemic chemotherapy with anthracycline#
* not eligible for autologous hematopoietic stem cell transplantation#
* at least one evaluable lesion#
* ECOG PS 0-1;
* 18-75 years; without other malignancy;
* proper functioning of the major organs.

Exclusion Criteria:

* double-hit lymphoma;
* previously received treatment of HDAC inhibitor;
* plan to receive autologous stem cell transplantation;
* involvement of central nervous system;
* previously received gemcitabine within the past 6 months;
* patients who received treatment for hematologic toxicity caused by previous chemotherapy within 7 days before enrollment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2023-03-11 (Actual)

PRIMARY OUTCOMES:
ORR | 4-years
  the proportion of patients who had CR, and PR according to the revised 2014 Lugano criteria for response assessment of lymphoma.

SECONDARY OUTCOMES:
DOR | 4-years
  the time from the first CR or PR to the first documented progressive disease (PD) or death, whichever occurred earlier.
PFS | 4-years
  the time from the date of enrollment until either PD or death.
OS | 4-years
  the time from the date of enrollment until death

OTHER OUTCOMES:
bio-marker analysis | 4-years
  Correlation between epigenetic factor mutation and efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zou Q, Zhang Y, Zhou H, Lai Y, Cao Y, Li Z, Su N, Li W, Huang H, Liu P, Ye X, Wu Y, Tan H, Zheng R, Wu B, Yang H, Zhong L, Lu Y, Liang Y, Sun P, Li L, Liu Y, Dai D, Xia Y, Cai Q. Chidamide, a Histone Deacetylase Inhibitor, Combined With R-GemOx in Relapsed/Refractory Diffuse Large B-Cell Lymphoma (TRUST): A Multicenter, Single-Arm, Phase 2 Trial. Cancer Med. 2025 May;14(9):e70919. doi: 10.1002/cam4.70919. PMID 40318003